CLINICAL TRIAL: NCT03730285
Title: Fast-track Discharge Combined With Treatment and Rehabilitation at Home With Telemedicine
Brief Title: Fast-track Discharge With Telemedicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Ole Winther Rasmussen, Senior Consultant, Kolding Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Fast-track telemedicine
Record Dates: First submitted 2016-02-28; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Emergencies
Keywords: telemedicine, patient satisfaction, randomization
MeSH Terms: conditions — Emergencies; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Active Comparator): Discharge with telemedicine contact to emergency nurse, doctor, and municipality
  Interventions: Device: Telemedicine
- Control (No Intervention): Standard care with 24-48 h observation at emergency unit

INTERVENTIONS:
Device: Telemedicine — Installation of videotelephone with broadband in patient's home
  Arms: Telemedicine

SUMMARY:
Evaluation of discharge after arrival at emergency unit, Kolding Hospital combined with treatment and rehabilitation in the home either by telemedicine or the usual treatment

DETAILED DESCRIPTION:
Participants are acute in-patients at the Medical Department, Kolding Hospital. Participants shall be informed about the project, and all screened initially within 30 minutes. After 3-4 hours adjusted treatment and possible need for new investigations are conducted. Patients are randomized at discharge to home treatment with rounds via telemedicine with support of emergency team of nurses or hospitalization in emergency unit. Observations, treatment and rehabilitation follow the same standards and guidelines for all patients. The cohort of patients is recruited between Oct 1, 2015 until January 1, 2016. The study is a randomized quality evaluation study of patient satisfaction, of the emergency team at Kolding Municipality, re-admittance rate, use of other health services, and new services from the municipality.

ELIGIBILITY:
Inclusion Criteria:

* municipal home care at admittance
* admitted to medical emergency care unit at Kolding Hospital

Exclusion Criteria:

* ketoacidosis,
* hyperosmolar diabetic coma,
* serious hypercalcemia,
* acute renal insufficiency with serum-creatinin > 175 mmol/l,
* serious cardiac failure
* septicemia
* acute coronary disease
* apoplexia cerebri
* neuroinfection
* progressive or active cancer
* hepatic disease
* serious psychiatric disease

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Walking distance | 3 months
  Measurement of walking distance regularly by home care nurse (in meters)

SECONDARY OUTCOMES:
Days of admittance | 3 months
  Days in hospital according t hospital charts
Fall in home | 3 months
  No. of falls in home recorded by home care nurse

CONTACTS AND LOCATIONS:
Overall Officials: Ole W Rasmussen, DrMedScie, Principal Investigator — Kolding Sygehs, Medical Department

IPD SHARING:
Plan to Share IPD: Yes
publication planned

REFERENCES:
- [Background] van Mastrigt GA, Joore MA, Nieman FH, Severens JL, Maessen JG. Health-related quality of life after fast-track treatment results from a randomized controlled clinical equivalence trial. Qual Life Res. 2010 Jun;19(5):631-42. doi: 10.1007/s11136-010-9625-5. Epub 2010 Mar 26. PMID 20340049
- [Background] Shea S, Weinstock RS, Teresi JA, Palmas W, Starren J, Cimino JJ, Lai AM, Field L, Morin PC, Goland R, Izquierdo RE, Ebner S, Silver S, Petkova E, Kong J, Eimicke JP; IDEATel Consortium. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus: 5 year results of the IDEATel study. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):446-56. doi: 10.1197/jamia.M3157. Epub 2009 Apr 23. PMID 19390093
- [Background] Mayes PA, Silvers A, Prendergast JJ. New direction for enhancing quality in diabetes care: utilizing telecommunications and paraprofessional outreach workers backed by an expert medical team. Telemed J E Health. 2010 Apr;16(3):358-63. doi: 10.1089/tmj.2009.0110. PMID 20406123